CLINICAL TRIAL: NCT01368666
Title: Perceval S Valve Clinical Trial for Extended CE Mark
Brief Title: Safety and Effectiveness Study of Perceval S Valve for Extended CE Mark
Acronym: CAVALIER
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: 5 years follow up completed in October 2018, long-term follow up terminated because of low data return
Sponsor: Corcym S.r.l (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TPS001
Record Dates: First submitted 2011-06-07; First posted 2011-06-08 (Estimated); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Aortic Valve Replacement
Keywords: Aortic valve replacement; Aortic stenosis; Biological valve; Sutureless valve; Stented valve; Aortic Valve Disease
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Perceval S Valve Prosthesis (Experimental): Patients who underwent replacement of diseased or malfunctioning native aortic valve with the Perceval S Valve prosthesis
  Interventions: Device: Perceval S Valve Prosthesis

INTERVENTIONS:
Device: Perceval S Valve Prosthesis — Replacement of diseased or malfunctioning native aortic valve with the Perceval S valve prosthesis

SUMMARY:
The primary objective of this clinical investigation is to assess the safety and effectiveness of the Perceval S valve at 12 months after implantation when used to replace a diseased or dysfunctional aortic valve or aortic valve prosthesis.

DETAILED DESCRIPTION:
Primary Endpoints

The primary endpoint of the clinical investigation is the evaluation of the safety and effectiveness of the Perceval S valve at 12 months after implant.

The safety of Perceval valve will be assessed in terms of percentage incidence of mortality and morbidity at 12 months after implant.

The effectiveness of the Perceval s valve will be assessed in terms of:

* Improvement of clinical status by mean of New York Heart Association (NYHA) functional class at 12 months after implant
* Haemodynamic performance through echocardiography parameters as mean gradient and peak gradient, effective orifice area (EOA), effective orifice area indexed (EOAI), performance index, cardiac output, cardiac index and degree of regurgitation at 12 months after implant

In order to determine mortality and morbidity, the following specific device related and procedure related adverse event categories will be assessed:

- valvular thrombosis, thromboembolism, hemorrhage (whether or not related to anti coagulant/ antiplatelet drug therapy) [all and major], paravalvular leak (all and major), endocarditis, hemolysis, structural valve deterioration, non structural dysfunction, reoperation (all and valve related), explant, death (all and valve related), device dislodgement and device migration

In order to assess the Haemodynamic performance the following echocardiography parameters will be measured:

- mean gradient and peak gradient, effective orifice area (EOA), effective orifice area indexed (EOAI), performance index, cardiac output, cardiac index and degree of regurgitation

Secondary Endpoints

The secondary endpoints of the clinical investigation are:

* Assessment of mortality and morbidity rates at discharge (or 30 days if the patient is still hospitalized) and at 3-6 months after implant
* Evaluation of the effectiveness of Perceval S valve in terms of improvement of clinical status assessed by means of NYHA functional class at discharge (or 30 days if the patient is still hospitalized), 3-6 months after surgery
* Evaluation of the effectiveness of Perceval S valve in terms of haemodynamic performance through echocardiography at discharge (or 30 days if the patient is still hospitalized) and 3-6 months after surgery
* Mortality and morbidity as well as haemodynamic parameters will be assessed

The Protocol has been amended (CAVALIER TPS001 Rev 4.0 Nov 17, 2017) to continue the follow up of a selection of implanted patients annually up to 10 years to evaluate long term device performance in the top enroller investigational sites.

The following secondary endpoints have been added:

* Assessment of mortality and morbidity rates annually until 10 years follow up. In order to determine mortality and morbidity, the following specific device related and procedure related adverse event categories will be assessed: valvular thrombosis, thromboembolism, hemorrhage (whether or not related to anti coagulant/ antiplatelet drug therapy) [all and major], paravalvular leak, endocarditis, hemolysis, structural valve deterioration, non structural dysfunction, reoperation, explant, death (all and valve related), device dislodgement and device migration.
* Evaluation of the effectiveness of Perceval valve in terms of improvement of clinical status assessed by NYHA change from baseline versus each follow-up up to 10 years.
* Evaluation of the effectiveness of Perceval valve in terms of haemodynamic performance through echocardiography at each follow up until 10 years. In order to assess the haemodynamic performance the following echocardiography parameters will be measured: mean gradient and peak gradient, effective orifice area (EOA), effective orifice area indexed (EOAI), performance index, cardiac output, cardiac index and degree of regurgitation.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects of age > 65 years;
2. Subjects with aortic valve stenosis or steno-insufficiency;
3. Subjects in which preoperative evaluation indicated the need for native or prosthetic aortic valve replacement with a biological prosthesis;
4. Subjects willing to sign the informed consent;
5. Subjects willing to undergo all medical follow-up, echocardiography examinations and laboratory tests planned for the Study

Exclusion Criteria:

1. Subjects involved in any other clinical study for drugs or devices;
2. Subjects with a previously implanted Perceval S prosthesis, within the clinical study, that requires replacement
3. Subjects with previous implantation of valve prostheses or annuloplasty ring not being replaced by the study valve
4. Subjects requiring simultaneous cardiac procedures, apart from septal myectomy and/or coronary by-pass
5. Subjects who require double or multiple valve replacement or repair in whom the mitral, tricuspid, or pulmonic valve would be replaced with a non-Perceval S valve or repaired
6. Subjects with aneurysmal dilation or dissection of the ascending aortic wall
7. Subjects needing non elective intervention
8. Subjects with active endocarditis
9. Subjects with active myocarditis
10. Subjects with congenital bicuspid aortic valve
11. Subjects with aortic root enlargement, where the ratio between the diameter of the sino-tubular junction and the annulus diameter, assessed by TTE, is > 1.3 (see Attachment 1 for reference)
12. Subjects with aortic root height (measured from aortic annulus to sino-tubular junction) ≥ 21 mm for size 21, ≥ 22.5 mm for size 23 and ≥ 24 mm for size 25, and ≥ 25 mm for size XL/27
13. Subjects with myocardial infarction < 90 days before the planned valve implant surgery
14. Subjects with known hypersensitivity to nickel alloys
15. The subject has a documented history of substance (drug or alcohol) abuse
16. The subject is a prison inmate, institutionalized, or is unable to give informed consent;
17. The subject has a major or progressive non-cardiac disease that, in the investigator's experience, results in a life expectancy shorter than 1 year, or the implant of the device produces an unacceptable increased risk to the patient
18. The subject is undergoing renal dialysis for chronic renal failure or has hyperparathyroidism
19. The subject has had an acute preoperative neurological deficit, myocardial infarction, or cardiac event that has not returned to baseline or stabilized ≥ 30 days prior to the planned valve implant surgery

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 658 (Actual)
Dates: Start 2010-02-23 (Actual); Primary Completion 2014-10-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of the safety: incidence of mortality | 12 months after OP
  Incidence of mortality
Evaluation of the safety: Incidence of morbidity | 12 months after OP
  Incidence of morbidity
  Mortality and morbidity, adverse event categories: valvular thrombosis, thromboembolism, hemorrhage, paravalvular leak, endocarditis, hemolysis, SVD, non structural dysfunction, reoperation, explant, death, device dislodgement and device migration
Evaluation of NYHA functional class | 12 months after OP
  Change of NYHA functional class
Evaluation of haemodynamic performance: mean and peak gradients | 12 months after OP
  Change of aortic mean gradient and peak gradient (mmHg)
Evaluation of haemodynamic performance: Effective Orifice Area (EOA) and Effective Orifice Area indexed (EOAI) | 12 months after OP
  Change of EOA (cm2) and EOAI (cm2/m2) PI, cardiac output, cardiac index and degree of regurgitation
Evaluation of haemodynamic performance: Cardiac Index | 12 months after OP
  Change of Cardiac Index (l/min/m2)
Evaluation of haemodynamic performance: Cardiac Output | 12 months after OP
  Change of Cardiac Output (l/min)
Evaluation of haemodynamic performance: incidence and degree of regurgitation | 12 months after OP
  Change of incidence (%) and degree of regurgitation (none, trace, mild, moderate, severe)

SECONDARY OUTCOMES:
Evaluation of the safety: incidence of mortality | 3-6 months
  Incidence of mortality
Evaluation of the safety: Incidence of morbidity | 3-6 months
  Incidence of morbidity
Evaluation of NYHA functional class | 3-6 months
  Change of NYHA functional class
Evaluation of haemodynamic performance | 3-6 months
  haemodynamic performance: mean gradient and peak gradient, EOA, EOAI, cardiac output, cardiac index and degree of regurgitation
Evaluation of the safety: Incidence of mortality | up to 10 years
  Incidence of mortality
Evaluation of the safety: Incidence of morbidity | up to 10 years
  Incidence of morbidity
Evaluation of NYHA functional class | up to 10 years
  Change of NYHA functional class
Evaluation of haemodynamic performance | up to 10 years
  haemodynamic performance: mean gradient and peak gradient, EOA, EOAI, cardiac output, cardiac index and degree of regurgitation

CONTACTS AND LOCATIONS:
Overall Officials: A. Haverich, Prof., Principal Investigator — Hannover Medical School
Locations (26):
- Austria (2):
  - Universitäts-Klinik für Chirurgie, Graz
  - Universitätsklinik für Chirurgie, Vienna
- Belgium (2):
  - Onze-Lieve-Vrouw (OLV) Ziekenhuis, Aalst
  - UZ Leuven, Leuven
- France (4):
  - CHRU de Lille, Lille
  - CHU - Nantes, Nantes
  - Institut Mutualiste Montsouris, Paris
  - Hôpital Cardiologique du Haut-Lévêque, Pessac
- Germany (12):
  - Herz- und Gefässzentrum Bad Bevensen, Bad Bevensen
  - RHÖN Klinikum AG, Herz- und Gefäß-Klinik GmbH, Bad Neustadt an der Saale
  - Herz- und Diabeteszentrum NRW, Bad Oeynhausen
  - Ruhr Universität Bochum, Bochum
  - Städtisches Klinikum Braunschweig, Braunschweig
  - Westdeutsches Herzzentrum, Essen
  - Universitäres Herzzentrum Hamburg GmbH, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Herzzentrum Leipzig, Leipzig
  - Deutsches Herzzentrum, Munich
  - Klinikum Nürnberg Süd, Nuremberg
  - Klinikum Oldenburg GmbH, Oldenburg
- Netherlands (3):
  - Academic Medical Center, Division of Cardio-thoracic Surgery, Amsterdam
  - Catharina Ziekenhuis, Eindhoven
  - St. Antonius Ziekenhuis, Nieuwegein
- Silesian Center for Heart Diseases, Zabrze, Poland
- Inselspital, Universitätsklinik für Herz- und Gefässchirurgie, Bern, Switzerland
- Genfield General Hospital, Leicester, United Kingdom

REFERENCES:
- [Result] Fischlein T, Meuris B, Folliguet T, Hakim-Meibodi K, Misfeld M, Carrel T, Zembala M, Cerutti E, Asch FM, Haverich A; CAVALIER Trial Investigators. Midterm outcomes with a sutureless aortic bioprosthesis in a prospective multicenter cohort study. J Thorac Cardiovasc Surg. 2022 Dec;164(6):1772-1780.e11. doi: 10.1016/j.jtcvs.2020.12.109. Epub 2021 Jan 13. PMID 33597099